CLINICAL TRIAL: NCT05356130
Title: Feasibility Pilot in Preparation for Large Pragmatic Encouragement Trial of Bright Light Therapy (BLT) for Depression
Brief Title: Bright Start Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Health Services Research
Other Study IDs: R34MH122550 (NIH); R34MH122550 (NIH)
Record Dates: First submitted 2022-04-20; First posted 2022-05-02 (Actual); Results first posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2024-09

CONDITIONS: Depression
Keywords: encouragement; coaching; adherence promotion; health education
MeSH Terms: conditions — Depression; Health Education

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment as Usual (TAU) (No Intervention): "Usual care services" control group
- Minimal BLT Encouragement (Active Comparator): Two minimal written communications promoting BLT as a promising treatment and outlining steps for patients to self-initiate. Arm 2 will not include any phone coaching or adherence promotion.
  Interventions: Behavioral: Written Educational Material on BLT
- Enhanced BLT Encouragement + Adherence Promotion (Active Comparator): 2-4 brief calls to encourage BLT use, advise on purchase of a light box (LB), assist with obtaining compensation for LB purchase, educate for correct LB use, and provide motivational interviewing (MI) as needed to promote adherence. Arm 3 participants will also receive the written educational material on BLT.
  Interventions: Behavioral: Written Educational Material on BLT; Behavioral: Enhanced BLT Encouragement and Adherence Promotion

INTERVENTIONS:
Behavioral: Written Educational Material on BLT — Participants in both Arms 2 and 3 will receive written information about how to obtain the greatest BLT benefit, including recommended day/time usage, session duration, eye distance from light box, the length of time to continue using, and the small risk of emergent mania or BD and how to recognize this. Written best practices for ideal BLT will be provided in both Arms 2 and 3 via secure EHR message, email, and/or USPS. PDFs of best practices for BLT will also be available for download on our study website.
  Arms: Enhanced BLT Encouragement + Adherence Promotion; Minimal BLT Encouragement
Behavioral: Enhanced BLT Encouragement and Adherence Promotion — BLT phone coaches will follow a four-step approach in engaging with Arm 3 participants: (a) provide encouragement to consider using BLT; (b) provide guidance regarding light box purchase and assist with obtaining compensation for purchase; (c) educate participants about ideal BLT use to obtain maximum benefit; and (d) provide ongoing brief telephonic adherence promotion and motivational interviewing (MI) where warranted to maximize persistent and appropriate BLT use.
  Arms: Enhanced BLT Encouragement + Adherence Promotion

SUMMARY:
The Bright Start study is a randomized trial to compare three approaches, or "arms", for delivering Bright Light Therapy (BLT) to real-world patients. Arm 1 participants will receive Kaiser Permanente (KP) treatment as usual (TAU) with no BLT assistance. Arm 2 participants will receive brief written educational material on BLT but no phone coaching. Arm 3 participants will receive written educational material and phone coaching assistance for BLT initiation and adherence. This pilot will prepare for a future, fully powered effectiveness trial and is not powered for hypothesis testing. Therefore, the investigators do not expect between-condition comparisons to yield significant differences. The investigators will conduct analyses similar to those that would be used in a subsequent fully powered trial of the same design. These pilot study analyses posit that (a) Arms 2+3 are superior to Arm 1 in PHQ-9 continuous depression response; and (b) Arm 3 is superior to Arm 2 in PHQ-9 continuous depression response. The investigators will also conduct exploratory analyses to prepare for a future fully powered trial.

DETAILED DESCRIPTION:
The most common treatments for depression are antidepressant medications (ADs) and psychotherapies such as cognitive behavioral therapy (CBT). However, these treatments yield only moderate benefits under ideal circumstances. These effects are further eroded when real world patients initiate treatments at low rates and have poor adherence or early discontinuation. This represents a depression care gap that supports the development and promotion of other interventions. One of these alternative treatments, bright light therapy (BLT), has established efficacy for seasonal affective disorder (SAD) and non-SAD depression, is relatively low cost, and has few adverse effects-but is often overlooked and has little presence in routine clinical care.

This R34 pilot study is in preparation for a subsequent large, pragmatic trial to examine the effectiveness of bright light therapy (BLT) for depression when delivered to real-world patients with little "scaffolding" typical of highly controlled efficacy trials. The investigators will conduct a feasibility pilot with a sample of 90 patients selected with a new clinical diagnosis of unipolar depression or SAD and PHQ-9 score >= 10, recorded in the health plan's electronic health record (EHR). Participants will be randomized to one of three arms:

* Arm 1 Treatment as Usual (TAU): A "usual care services" control group (e.g., ADs, psychotherapy; all TAU is permitted and will be recorded for all participants in all conditions);
* Arm 2 TAU + Minimal BLT Encouragement: TAU plus two minimal written communications (mailed letter, secure EHR message, or email) promoting BLT as a promising treatment and outlining steps for patients to self-initiate; Arm 2 will not include any phone coaching or adherence promotion;
* Arm 3 TAU + Enhanced BLT Encouragement + Adherence Promotion: TAU plus 2-4 brief calls to encourage BLT use, advise on purchase of a light box (LB), assist with obtaining compensation for LB purchase, educate for correct LB use, and provide motivational interviewing (MI) as needed to promote adherence.

The primary outcome is PHQ-9 self-reported depression symptoms; the primary test of BLT effectiveness is the contrast between Arms 2+3 vs. Arm 1. This underpowered pilot study is not powered for hypothesis testing. Therefore, the investigators do not expect between-condition comparisons to yield significant differences. Nonetheless, as part of this pilot the investigators will conduct analyses similar to those that would be used in the planned, subsequent fully powered trial of the same design. These pilot-study analyses posit that (a) Arms 2+3 are superior to Arm 1 in PHQ-9 continuous depression response; and (b) Arm 3 is superior to Arm 2 in PHQ-9 continuous depression response. The investigators will conduct exploratory analyses to prepare for a future fully powered trial. The investigators will examine other secondary outcomes including anxiety, disability, and mood seasonality, and other secondary contrasts; e.g., Arm 2 vs Arm 3. The investigators will also examine moderation effects; variation of BLT effects in subgroups (e.g., those receiving vs. not receiving TAU antidepressants); and the investigators will examine mechanisms of BLT and MI intervention effects via candidate mediators including normalized circadian rhythm, improved sleep, and increased physical activity (for BLT), and readiness for change (for MI). This pilot will yield feasibility products to assist with successful conduct of a subsequent full trial: estimates of recruitment success, participant retention, and adherence with BLT protocol; refinement of the adherence promotion protocol; and an estimate (with wide confidence intervals) of BLT effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-69 years, inclusive
* New episode of unipolar depression within the last month, defined as: New ICD-10 diagnosis of SAD or unipolar depression (i.e., major depression, minor depression, depression not otherwise specified, and/or adjustment disorder with depressed mood) AND usual care administration of the PHQ-9 depression scale in the last 30 days, with a total score of 10 or higher
* Participant must have a kp.org MyChart account, with evidence of use in the last 12 months
* Able and willing to conduct study assessments and phone coaching in English
* Phone and internet access

Exclusion Criteria:

* Chronic depression: ICD-10 diagnosis of SAD or unipolar depression in the 6 months prior to case-identification
* Elevated PHQ-9 (score of 10 or higher) in the 6 months prior to case identification
* Active electronic health record (EHR) diagnoses and prescriptions representing any of the following contraindications for BLT: Conditions that might render skin or eyes more vulnerable to phototoxicity (e.g., ophthalmic disorders such as cataract, macular degeneration, glaucoma, retinitis pigmentosa; disorders affecting the retina such as retinopathy, diabetes, herpes); or photosensitive skin; or if they are taking a photosensitizing medication or herb (e.g., St. John's wort or a psoralen)
* EHR-recorded diagnoses of bipolar disorder I or II
* Participation barriers (e.g., terminal end-stage cancer, moving out of the region, no locator information)
* Contraindicated diagnoses or medications (see EHR exclusion criteria above) in case these are known to patients but are not EHR-recorded (e.g., if they were diagnosed with a contraindicated condition before becoming a KP member and have not yet sought care for it)
* Contraindicated diagnoses or medications (see EHR exclusion criteria) newly reported that were not captured in the EHR
* Emergent bipolar, manic, mixed symptoms that may not have been formally diagnosed yet (e.g., significant mood swings, excessive increases in energy, dramatically less need for sleep)

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2022-02-17 (Actual); Primary Completion 2023-08-20 (Actual); Study Completion 2024-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Greg Clarke, PhD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Northwest Center for Health Research, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment as Usual (TAU) | Minimal BLT Encouragement | Enhanced BLT Encouragement + Adherence Promotion
Started | 31 | 30 | 31
Completed | 31 | 30 | 28
Not Completed | 0 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment as Usual (TAU) | Minimal BLT Encouragement | Enhanced BLT Encouragement + Adherence Promotion | Total
Number analyzed (Participants) | 31 | 30 | 31 | 92
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 31 | 30 | 31 | 92
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.5 (9.9) | 34.3 (9.5) | 37.0 (9.5) | 35.6 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 18 | 21 | 60
  Male | 10 | 12 | 10 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 7 | 17
  Not Hispanic or Latino | 26 | 25 | 24 | 75
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 0 | 0 | 0 | 0
  White | 22 | 21 | 22 | 65
  More than one race | 6 | 6 | 7 | 19
  Unknown or Not Reported | 0 | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Patient Health Questionnaire-9 (PHQ-9)
Description: Change on continuous total score of the PHQ-9, a measure of self-reported depression symptoms. Minimum score = 0, maximum score = 27, higher scores = worse outcome.
Time Frame: Baseline through follow-up at 2, 4 and 6 months post-enrollment
Population: Even though everyone contributes to the statistical analysis, we only report means for those people with observed values.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment as Usual (TAU) | Minimal BLT Encouragement | Enhanced BLT Encouragement + Adherence Promotion
Number analyzed (Participants) | 31 | 30 | 31
score on a scale
  Baseline: number analyzed (Participants) | 31 | 29 | 31
  Baseline | 12.9 (5.3) | 13.7 (5.1) | 13.8 (6.0)
  2-Month Follow-up: number analyzed (Participants) | 27 | 27 | 25
  2-Month Follow-up | 12.2 (5.6) | 10.8 (6.5) | 9.3 (5.3)
  4-Month Follow-up: number analyzed (Participants) | 25 | 26 | 21
  4-Month Follow-up | 10.0 (4.8) | 10.0 (5.7) | 9.1 (5.2)
  6-Month Follow-up: number analyzed (Participants) | 27 | 27 | 20
  6-Month Follow-up | 10.4 (6.1) | 9.4 (5.4) | 8.3 (6.2)

2. Secondary Outcome: Quick Inventory of Depressive Symptomatology, Self-report (QIDS-SR)
Description: Change on the QIDS-SR, a self-reported measure of depression symptoms. Minimum score = 0, maximum score = 48, where higher scores = worse outcome.
Time Frame: Baseline through follow-up at 2, 4 and 6 months post-enrollment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment as Usual (TAU) | Minimal BLT Encouragement | Enhanced BLT Encouragement + Adherence Promotion
Number analyzed (Participants) | 31 | 30 | 31
score on a scale
  Baseline: number analyzed (Participants) | 26 | 30 | 30
  Baseline | 13.2 (5.1) | 13.2 (4.0) | 12.2 (4.8)
  2-Month Follow-up: number analyzed (Participants) | 23 | 26 | 25
  2-Month Follow-up | 11.8 (4.0) | 11.3 (4.6) | 9.7 (5.3)
  4-Month Follow-up: number analyzed (Participants) | 23 | 25 | 21
  4-Month Follow-up | 9.7 (5.1) | 9.9 (4.3) | 8.9 (4.1)
  6-Month Follow-up: number analyzed (Participants) | 22 | 26 | 19
  6-Month Follow-up | 10.0 (4.8) | 10.0 (4.5) | 8.8 (5.6)

3. Secondary Outcome: Pittsburgh Sleep Quality Index (PSQI)
Description: Change on self-rated PSQI questionnaire to assess sleep quality and disturbances. Minimum score = 0, maximum score = 21, where higher scores = worse outcome.
Time Frame: Baseline through follow-up at 2, 4 and 6 months post-enrollment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment as Usual (TAU) | Minimal BLT Encouragement | Enhanced BLT Encouragement + Adherence Promotion
Number analyzed (Participants) | 31 | 30 | 31
score on a scale
  Baseline | 9.6 (3.4) | 9.0 (3.5) | 9.1 (3.8)
  2-Month Follow-up: number analyzed (Participants) | 27 | 26 | 26
  2-Month Follow-up | 10.1 (3.8) | 8.0 (3.1) | 8.0 (3.4)
  4-Month Follow-up: number analyzed (Participants) | 26 | 26 | 21
  4-Month Follow-up | 9.4 (4.2) | 7.5 (3.3) | 7.1 (2.8)
  6-Month Follow-up: number analyzed (Participants) | 27 | 27 | 20
  6-Month Follow-up | 9.3 (4.0) | 7.2 (2.8) | 7.1 (3.5)
Statistical Analysis 1: Comparison: Treatment as Usual (TAU) vs Minimal BLT Encouragement vs Enhanced BLT Encouragement + Adherence Promotion; We conducted the same two independent planned comparisons: "Enhanced BLT Encouragement + Adherence Promotion" compared to "Minimal BLT Encouragement"; "Minimal BLT Encouragement" and "Enhanced BLT Encouragement + Adherence Promotion" compared to "TAU"; Test type: Superiority; p = 0.014, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 6 months
Arm/Group | Treatment as Usual (TAU) | Minimal BLT Encouragement | Enhanced BLT Encouragement + Adherence Promotion
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/30 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/30 | 0/31
Other Adverse Events (participants affected / at risk) | 0/31 | 0/30 | 0/31

LIMITATIONS AND CAVEATS:
The relatively small pilot sample size was planned from the beginning to be insufficient for fully powered hypothesis testing, but sufficient for protocol/procedures feasibility testing. Effect sizes should be interpreted with caution.

The racial and ethnic makeup of the sample limits the generalizability of results.

We intentionally enrolled either SAD or non-SAD depression, which may limit generalizability due to durable medical equipment reimbursement only available for SAD depression.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2023-09-13): https://cdn.clinicaltrials.gov/large-docs/30/NCT05356130/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-02): https://cdn.clinicaltrials.gov/large-docs/30/NCT05356130/SAP_001.pdf
  • Informed Consent Form (2022-06-09): https://cdn.clinicaltrials.gov/large-docs/30/NCT05356130/ICF_002.pdf